CLINICAL TRIAL: NCT00108485
Title: Randomized, Double-blind, Placebo-controlled Trial of Niaspan® in Patients With Overt Diabetic Nephropathy and Moderate Renal Impairment
Brief Title: Study of the Use of Niaspan for Treatment of Dyslipidemia in Diabetic Nephropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit sufficient study subjects
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ronald Goldberg, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20043224
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 2; Kidney Failure, Chronic; Hyperlipidemia
Keywords: Diabetes Mellitus, Type 2; Kidney Failure, Chronic; Hyperlipidemia; Randomized Controlled Trials
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic; Hyperlipidemias | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended release niacin (Active Comparator): Extended release niacin 1500-2000 mg daily versus placebo comparator
  Interventions: Drug: Extended release niacin
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Extended release niacin — Extended release niacin 1500-2000mg once daily
  Other Names: Niaspan
  Arms: Extended release niacin
Other: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to test the effectiveness and tolerability of Niaspan® to improve the levels of blood fats ("good" and "bad" cholesterol and triglyceride levels) in people who have kidney damage due to diabetes. A secondary goal is to test whether Niaspan® slows down further development of kidney damage.

DETAILED DESCRIPTION:
Diabetic nephropathy is the leading cause of end stage kidney disease in the United States. Patients with chronic kidney disease have a markedly increased risk of death from cardiovascular disease, and traditional risk factors such as hyperlipidemia have been shown to be of critical importance. Almost 90% of patients with diabetes and chronic kidney disease have lipid abnormalities. Here, we investigate whether Niaspan, taken in addition to lipid-lowering drugs referred to as "statins", will decrease LDL cholesterol and increase LDL particle size, increase HDL, reduce proteinuria, and reduce the speed of loss of renal function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Diagnosis of chronic kidney disease stage 2 or 3 with an estimated GFR of 30-89 ml/min using the four variable MDRD (Modification of Diet in Renal Disease Study Group) formula
* Presence of microalbuminuria or proteinuria less than 3.5 g/d
* Diagnosis of hyperlipidemia currently treated with a "statin" drug

Exclusion Criteria:

* Not meeting inclusion criteria
* HDL-C > 40 mg/dL for men, > 50 mg/dL for women
* TG (triglycerides) < 150 mg/dL and > 800 mg/dL
* Documented intolerance to Niaspan or Aspirin
* Treatment with other lipid-lowering agents (fibrates, BAS [bile acid sequestrants], or ezetimibe)
* Elevated transaminases (AST or ALT >1.3 x ULN)
* Unstable type 2 diabetes (FBG >200 mg/dL or HbA1c >9.5%)
* Known seropositivity for Hepatitis B, C, or HIV
* Documented history of malignancy
* Age < 18 years
* Pregnant women or nursing mothers
* Inability to give informed consent
* Start or change in "statin" dose < 2 months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldberg, MD, Principal Investigator — University of Miami, Miami, FL
Locations (1):
- Univesity of Miami/Diabetes Research Institute, Miami, Florida, United States

REFERENCES:
- [Background] Grundy SM, Vega GL, McGovern ME, Tulloch BR, Kendall DM, Fitz-Patrick D, Ganda OP, Rosenson RS, Buse JB, Robertson DD, Sheehan JP; Diabetes Multicenter Research Group. Efficacy, safety, and tolerability of once-daily niacin for the treatment of dyslipidemia associated with type 2 diabetes: results of the assessment of diabetes control and evaluation of the efficacy of niaspan trial. Arch Intern Med. 2002 Jul 22;162(14):1568-76. doi: 10.1001/archinte.162.14.1568. PMID 12123399
- [Background] Wolfe ML, Vartanian SF, Ross JL, Bansavich LL, Mohler ER 3rd, Meagher E, Friedrich CA, Rader DJ. Safety and effectiveness of Niaspan when added sequentially to a statin for treatment of dyslipidemia. Am J Cardiol. 2001 Feb 15;87(4):476-9, A7. doi: 10.1016/s0002-9149(00)01410-7. PMID 11179541
- [Background] Guyton JR, Blazing MA, Hagar J, Kashyap ML, Knopp RH, McKenney JM, Nash DT, Nash SD. Extended-release niacin vs gemfibrozil for the treatment of low levels of high-density lipoprotein cholesterol. Niaspan-Gemfibrozil Study Group. Arch Intern Med. 2000 Apr 24;160(8):1177-84. doi: 10.1001/archinte.160.8.1177. PMID 10789612
- [Background] Whitney EJ, Krasuski RA, Personius BE, Michalek JE, Maranian AM, Kolasa MW, Monick E, Brown BG, Gotto AM Jr. A randomized trial of a strategy for increasing high-density lipoprotein cholesterol levels: effects on progression of coronary heart disease and clinical events. Ann Intern Med. 2005 Jan 18;142(2):95-104. doi: 10.7326/0003-4819-142-2-200501180-00008. PMID 15657157
- [Background] Owada A, Suda S, Hata T. Antiproteinuric effect of niceritrol, a nicotinic acid derivative, in chronic renal disease with hyperlipidemia: a randomized trial. Am J Med. 2003 Apr 1;114(5):347-53. doi: 10.1016/s0002-9343(02)01567-x. PMID 12714122

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended Release Niacin | Placebo
Started | 5 | 4
Completed | 2 | 2
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Release Niacin | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Proteinuria
Time Frame: Baseline, 1 year
Population: Nine participants were enrolled into this study, however baseline data is only available for 2 participants (1 from the Extended Release Niacin arm and 1 from the Placebo arm). Data was only analyzed for 2 participants.
Measure: Number; unit: mg/dL
Arm/Group | Extended Release Niacin | Placebo
Number analyzed (Participants) | 1 | 1
mg/dL | 42 | 63

ADVERSE EVENTS:
Description: Solicited by questionnaire.
Arm/Group | Extended Release Niacin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/5 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Niacin (N=5) | Placebo (N=4)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Subpleural Nodule (Vascular disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bilateral Calf Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Itching Upper Extremeties (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back and Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leg Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of study lead to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No